CLINICAL TRIAL: NCT07281235
Title: Perioperative Analgesia With Ultrasound Guided Erector Spinae Block Versus Ultrasound Guided Caudal Block in Children
Brief Title: Perioperative Analgesia Using Ultrasound Guided Erector Spinae Block vs Ultrasound Guided Caudal Block for Pain Control in Children Aged 2-7 Years Undergoing Lower Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 9250511
Record Dates: First submitted 2025-11-13; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2024-12

CONDITIONS: Local Analgesia Via Infiltration; Caudal Epidural Anesthesia; Caudal Block; Caudal Block for Postoperative Analgesia; Caudal Anesthesia; Erector Spinae Plane Block; Children
Keywords: Erector Spinae Block; Caudal Block; Pediatrics; llower abdominal surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal Block Group (Active Comparator): Patients who received ultrasound guided Caudal Block
  Interventions: Procedure: Caudal Block Anesthesia
- Erector Spinae Plane Block Group (Active Comparator): Patients who received ultrasound guided Erector Spinae Block
  Interventions: Procedure: Ultrasound Guided Bilateral single shot Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Ultrasound Guided Bilateral single shot Erector Spinae Plane Block — Ultrasound Guided Erector Spinae Plane block given bilaterally at level of L1.
  Other Names: Ultrasound Guided erector spinae pkane block
  Arms: Erector Spinae Plane Block Group
Procedure: Caudal Block Anesthesia — Ukltrasound Guided Caudal Epidural Block
  Arms: Caudal Block Group

SUMMARY:
The goal of this prospective study is to is to evaluate the perioperative pain management of Erector Spinae Block versus Caudal Block using the Face, Legs, Activity, Cry, Conceal ability (FLACC) Pain Scale inn children aged 2 to 7 years old. The main question it aims to answer is:

Which block is more efficient in the perioperative period?

Participants will be evaluated intraoperative and postoperative for hemodynamic changes and their pain will evaluated according to the FLACC score.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2-7 years old.
* ASA I-II.
* Elective surgery under general anaesthesia.
* Lower abdominal surgery.

Exclusion Criteria:

* Parent/caregiver refusal.
* Allergy to one of the study medications.
* Renal or cardiac disease.
* Infection or redness at the site of injection.
* Clinically significant coagulopathy.
* Spinal anomalies.
* Altered mental status.
* Developmental delay.
* Additional surgery at different surgical sites.
* Block failure.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of postoperative pain management of Erector Spinae Block versus Caudal Block. | At 15 minutes and 30 minutes in PACU, then every 2 hours up to 8 hours after surgery.
  Evaluate postoperative pain using the Face, Legs, Activity, Cry, Consolability (FLACC) scale.
  A score of 0 = no pain, 10 = severe pain. A score ≥4 requires rescue analgesia.

SECONDARY OUTCOMES:
Changes to heart rate (beats/minute) | T0: before induction of anesthesia T1: after induction of anesthesia (within 5 minutes) T2: immediately after block placement (within 5 minutes) T3: start of surgery T4: every 10 minutes intraoperative until the end of surgery T5: end of surgery
  Changes to heart rate (beats/minute) recorded before surgery, during surgery and immediately after surgery
The time to first rescue analgesic. | from 0 to 8 hours after block administration
  Time from block administration to the patient's first requirement for rescue analgesia.
Total postoperative analgesic requirements. | from 0 to 8 hours after block administration
  Amount and frequency of analgesia patient requested
Parent satisfaction with a 5-point Likert scale questionnaire. | At 8 hours after block administration
  Parent or caregiver satisfaction about block efficiency on a scale of 1 to 5.
Number of patients required rescue analgesic postoperatively. | From 0 to 8 hours after surgery.
  Number of patiebts of asked for rescue analgesia is recorded.
Time to Modified Aldrete score ≥9. | from arrival to PACU (0 hours) until achieving an Aldrete score ≥9 (expected within 60 minutes)
  Postoperative recovery was assessed using the Modified Aldrete Scoring System, which evaluates five physiological criteria: activity, respiration, circulation, consciousness, and oxygen saturation
Incidence of any adverse effects. | from end of surgery (0 hours) to 8 hours postoperatively
  Any side effects reported by the patient related to analgesia.
Changes to mean arterial pressure (MAP) | T0: before induction of anesthesia T1: after induction of anesthesia (within 5 minutes) T2: immediately after block placement (within 5 minutes) T3: start of surgery T4: every 10 minutes intraoperative until the end of surgery T5: end of surgery
  changes to mean arterial pressure (MAP) (mmHg) before surgery, during surgery and immediately after surgey
Changes to oxygen saturation | T0: before induction of anesthesia T1: after induction of anesthesia (within 5 minutes) T2: immediately after block placement (within 5 minutes) T3: start of surgery T4: every 10 minutes intraoperative until the end of surgery T5: end of surgery
  Changes to oxygen saturation before surgery, during surgery and immediately after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf A Abdelhalim, Doctorate, Study Chair — Professor of Anesethia and Surgical Intensive Care.; Ahmed M El Attar, Doctorate, Study Director — Professor of Anesethia and Surgical Intensive Care.; Aliaa R Abdel Aziz, Doctorate, Study Director — Assistant Professor of Anesethia and Surgical Intensive Care.
Locations (1):
- El Shatby University Hospital for Children, Alexandria, EL Shatby, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aksu C, Gurkan Y. Defining the Indications and Levels of Erector Spinae Plane Block in Pediatric Patients: A Retrospective Study of Our Current Experience. Cureus. 2019 Aug 8;11(8):e5348. doi: 10.7759/cureus.5348. PMID 31602352
- [Background] Aldrete JA. The post-anesthesia recovery score revisited. J Clin Anesth. 1995 Feb;7(1):89-91. doi: 10.1016/0952-8180(94)00001-k. No abstract available. PMID 7772368
- [Background] Chanthong P, Abrishami A, Wong J, Herrera F, Chung F. Systematic review of questionnaires measuring patient satisfaction in ambulatory anesthesia. Anesthesiology. 2009 May;110(5):1061-7. doi: 10.1097/ALN.0b013e31819db079. PMID 19352161
- [Background] Lucente M, Ragonesi G, Sanguigni M, Sbaraglia F, Vergari A, Lamacchia R, Del Prete D, Rossi M. Erector spinae plane block in children: a narrative review. Korean J Anesthesiol. 2022 Dec;75(6):473-486. doi: 10.4097/kja.22279. Epub 2022 Jul 5. PMID 35790215
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Kollipara N, Kodali VRK, Parameswari A. A randomized double-blinded controlled trial comparing ultrasound-guided versus conventional injection for caudal block in children undergoing infra-umbilical surgeries. J Anaesthesiol Clin Pharmacol. 2021 Apr-Jun;37(2):249-254. doi: 10.4103/joacp.JOACP_361_19. Epub 2021 Jul 15. PMID 34349375
- [Background] Chen CP, Lew HL, Tang SF. Ultrasound-guided caudal epidural injection technique. Am J Phys Med Rehabil. 2015 Jan;94(1):82-4. doi: 10.1097/PHM.0000000000000047. No abstract available. PMID 24722013
- [Background] Opfermann P, Kraft F, Obradovic M, Zadrazil M, Schmid W, Marhofer P. Ultrasound-guided caudal blockade and sedation for paediatric surgery: a retrospective cohort study. Anaesthesia. 2022 Jul;77(7):785-794. doi: 10.1111/anae.15738. Epub 2022 Apr 22. PMID 35460068
- [Background] Kao SC, Lin CS. Caudal Epidural Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:9217145. doi: 10.1155/2017/9217145. Epub 2017 Feb 26. PMID 28337460
- [Background] Lamontagne LL, Hepworth JT, Salisbury MH. Anxiety and postoperative pain in children who undergo major orthopedic surgery. Appl Nurs Res. 2001 Aug;14(3):119-24. doi: 10.1053/apnr.2001.24410. PMID 11481590
- [Background] Victoria NC, Murphy AZ. Exposure to Early Life Pain: Long Term Consequences and Contributing Mechanisms. Curr Opin Behav Sci. 2016 Feb;7:61-68. doi: 10.1016/j.cobeha.2015.11.015. PMID 27525299
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Gehdoo Rp. Post operative pain management in paediatric patients. IndianJ Anaesth 2004; 48(5):406-14.
- [Background] Smith HA, Berutti T, Brink E, Strohler B, Fuchs DC, Ely EW, Pandharipande PP. Pediatric critical care perceptions on analgesia, sedation, and delirium. Semin Respir Crit Care Med. 2013 Apr;34(2):244-61. doi: 10.1055/s-0033-1342987. Epub 2013 May 28. PMID 23716315
- [Background] Birnie KA, Noel M, Chambers CT, Uman LS, Parker JA. Psychological interventions for needle-related procedural pain and distress in children and adolescents. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005179. doi: 10.1002/14651858.CD005179.pub4. PMID 30284240
- [Background] Ingelmo P, Rivera G, Baird R. Pain control after pediatric surgery: learning from the past to perfect the future. Pain Manag. 2016;6(1):9-12. doi: 10.2217/pmt.15.51. Epub 2015 Dec 17. No abstract available. PMID 26677915
- [Result] Abdelrazik AN, Ibrahim IT, Farghaly AE, Mohamed SR. Ultrasound-guided Erector Spinae Muscle Block Versus Ultrasound-guided Caudal Block in Pediatric Patients Undergoing Lower Abdominal Surgeries. Pain Physician. 2022 Jul;25(4):E571-E580. PMID 35793181

DOCUMENTS (1):
  • Study Protocol (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT07281235/Prot_000.pdf